CLINICAL TRIAL: NCT01345227
Title: Pilot Study to Assess Feasibility and Safety of Bone Marrow as Alternative Site in Islet Transplant Patients
Brief Title: Bone Marrow as an Alternative Site for Islet Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ospedale San Raffaele (Other)
Collaborators: European Union (Other)
Responsible Party: Principal Investigator, Piemonti Lorenzo, Director Islet Transplantation Program, Ospedale San Raffaele
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BMT1
Record Dates: First submitted 2011-04-28; First posted 2011-05-02 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2012-10

CONDITIONS: Type 1 Diabetes; Postpancreatectomy Hyperglycemia
Keywords: Type 1 diabetes; islet transplantation; autotransplantation
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intra BM islet infusion (Experimental): single intra BM islet infusion at the level of the iliac crest will be performed in patients having contraindications for intraportal infusion
  Interventions: Procedure: Intra bone marrow islet infusion

INTERVENTIONS:
Procedure: Intra bone marrow islet infusion — A needle for bone marrow aspiration (14 G) will be inserted into the superior-posterior iliac crest and islet suspension (1:2.5; tissue:Ringer's Lactate solution) will be infused. The entire intraBM-injection procedure last 8-15 min from the beginning of anaesthesia (short propofol sedation).

SUMMARY:
The goal of this study is to evaluate safety and feasibility of bone marrow (BM) as site for islet transplantation (Tx) in humans. The investigators hypothesis is that BM represents a better site than liver thanks to its potential capacity to favor islet engraftment in face of a more easiness of access and bioptic follow up.

DETAILED DESCRIPTION:
We were permitted to perform single intra BM islet infusion at the level of the iliac crest in patients having contraindications for intraportal infusion. A needle for BM aspiration (14 G) is inserted into the superior-posterior iliac crest and islet suspension (1:2.5; tissue:Ringer's Lactate solution) is infused. The entire intraBM-injection procedure lasted 8-15 min from the beginning of anaesthesia (short propofol sedation).

ELIGIBILITY:
Inclusion Criteria:

* diabetic patients eligible for pancreatic islet transplantation based on local accepted practice and guidelines. This includes at least: a)clinical history compatible with T1D with insulin-dependence for >5 years; b) undetectable stimulated (arginine or MMTT) C-peptide levels (<0.3 ng/mL) in the 12 months before transplant c)presence of severe hypoglycaemic events
* patients undergoing total pancreatectomy because of anastomosis leakage after pancreatoduodenectomy or because of pancreatic anastomosis is made impracticable by technical difficulties and/or high risk of leakage.
* presence of contraindications for intraportal islet infusion

Exclusion Criteria:

* presence of hematologic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2009-08; Primary Completion 2011-04 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Adverse events related to the procedure of intra bone marrow islet infusion | up to 3 years

SECONDARY OUTCOMES:
Beta-cell function | up to 3 years
  Beta-cell function will be assessed by fasting C peptide, HbA1c,glycaemia, change in average daily insulin requirements, basal (fasting) and -10 to 120 min time course of glucose, C-peptide and insulin derived from the arginine test, beta-score and Transplant Estimated Function

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Piemonti, MD, Principal Investigator — Fondazione Centro San Raffaele del Monte Tabor; Paola Maffi, MD, Study Director — Fondazione Centro San Raffaele del Monte Tabor
Locations (1):
- IRCCS San Raffaele, Milan, Italy

REFERENCES:
- [Background] Cantarelli E, Melzi R, Mercalli A, Sordi V, Ferrari G, Lederer CW, Mrak E, Rubinacci A, Ponzoni M, Sitia G, Guidotti LG, Bonifacio E, Piemonti L. Bone marrow as an alternative site for islet transplantation. Blood. 2009 Nov 12;114(20):4566-74. doi: 10.1182/blood-2009-03-209973. Epub 2009 Sep 22. PMID 19773545
- [Background] Ciceri F, Piemonti L. Bone marrow and pancreatic islets: an old story with new perspectives. Cell Transplant. 2010;19(12):1511-22. doi: 10.3727/096368910X514279. Epub 2010 Aug 17. PMID 20719074
- [Result] Maffi P, Balzano G, Ponzoni M, Nano R, Sordi V, Melzi R, Mercalli A, Scavini M, Esposito A, Peccatori J, Cantarelli E, Messina C, Bernardi M, Del Maschio A, Staudacher C, Doglioni C, Ciceri F, Secchi A, Piemonti L. Autologous pancreatic islet transplantation in human bone marrow. Diabetes. 2013 Oct;62(10):3523-31. doi: 10.2337/db13-0465. Epub 2013 Jun 3. PMID 23733196
- [Derived] Maffi P, Nano R, Monti P, Melzi R, Sordi V, Mercalli A, Pellegrini S, Ponzoni M, Peccatori J, Messina C, Nocco A, Cardillo M, Scavini M, Magistretti P, Doglioni C, Ciceri F, Bloem SJ, Roep BO, Secchi A, Piemonti L. Islet Allotransplantation in the Bone Marrow of Patients With Type 1 Diabetes: A Pilot Randomized Trial. Transplantation. 2019 Apr;103(4):839-851. doi: 10.1097/TP.0000000000002416. PMID 30130323